CLINICAL TRIAL: NCT01835236
Title: A Randomized Phase II Trial of Pertuzumab in Combination With Trastuzumab With or Without Chemotherapy, Both Followed by T-DM1 in Case of Progression, in Patients With HER2-positive Metastatic Breast Cancer
Brief Title: Trastuzumab & Pertuzumab Followed by T-DM1 in MBC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 22/10; 2012-002556-17 (EudraCT Number); UNICANCER UC-0140/1207 (Other: Unicancer)
Record Dates: First submitted 2013-04-15; First posted 2013-04-18 (Estimated); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast cancer; HER2-positive; Metastases
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Trastuzumab; pertuzumab; Paclitaxel; Vinorelbine; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trastuzumab, Pertuzumab, T-DM1 (Active Comparator): First line therapy: Trastuzumab, Pertuzumab Second line therapy: T-DM1
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: T-DM1
- Trastuzumab, Pertuzumab, Paclitaxel or Vinorelbine plus T-DM1 (Active Comparator): First line therapy: Trastuzumab, Pertuzumab, Paclitaxel or Vinorelbine Second line therapy: T-DM1
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Paclitaxel; Drug: Vinorelbine; Drug: T-DM1

INTERVENTIONS:
Drug: Trastuzumab — First administration (loading dose) 8 mg/kg i.v. infusion over 90 min.
  - then every 3 weeks until progression 6 mg/kg i.v. infusion over 30 to 90 min.
  Other Names: Herceptin
Drug: Pertuzumab — First administration (loading dose) 840 mg i.v. infusion over 60 min.
  - then every 3 weeks until progression 420 mg i.v. infusion over 30 to 60 min.
  Other Names: Perjeta
Drug: Paclitaxel — Day 1, 8 and 15; every 4 weeks for ≥4 months 90 mg/m2 i.v. infusion
  Other Names: Taxol
  Arms: Trastuzumab, Pertuzumab, Paclitaxel or Vinorelbine plus T-DM1
Drug: Vinorelbine — First administration: Day 1 and 8 25 mg/m2 i.v. infusion
  * then day 1 and 8, every 3 weeks for ≥4 months 30 mg/m2 i.v. infusion
  Other Names: Navelbine
  Arms: Trastuzumab, Pertuzumab, Paclitaxel or Vinorelbine plus T-DM1
Drug: T-DM1 — Every 3 weeks until unacceptable toxicity or progressive disease is observed 3.6 mg/kg i.v. infusion First dose: over 90 min (± 10 min.) Subsequent doses: over 30 min. (± 10 min.)
  Other Names: Trastuzumab emtansine

SUMMARY:
In HER2-positive metastatic breast cancer, trastuzumab based treatment is the standard of care as long as there are no contraindications to trastuzumab. Frequently, trastuzumab is being combined with taxanes in the first-line setting. However, since therapy with trastuzumab is active even in the absence of chemotherapy in HER2-positive MBC, the optimal treatment strategy either in combination or in sequence with chemotherapy is still under debate. This randomized phase II trial is studying a new strategy for the treatment of metastatic breast cancer with HER2-positive. First-line treatment consists of trastuzumab and pertuzumab, a treatment without chemotherapy. In case of disease progression, chemotherapy with T-DM1 is then performed as second-line treatment. Third-line and further line therapies are performed according to the physician's discretion. If this new therapeutic strategy is as effective and better tolerated than the conventional strategy, this would mean a serious breakthrough in the treatment of HER2-positive metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

-To evaluate the efficacy in terms of overall survival (OS) at 24 months of a chemotherapy-free dual HER2-inhibition with trastuzumab and pertuzumab (first-line) followed by T-DM1 (second-line) and of a chemotherapy-containing dual HER2-inhibition with trastuzumab and pertuzumab (first-line) followed by T-DM1 (second-line) in patients with HER2-positive metastatic breast cancer.

Secondary

* To evaluate other efficacy parameter
* To evaluate the safety and tolerability profile of the two treatment strategies
* To evaluate the Quality of Life (QoL)
* To learn how patients are treated after trial treatment

OUTLINE: This is a multicenter study. Patients are stratified according to hormone receptor status (positive vs negative), prior trastuzumab (never or >12 months vs ≤12 months after last infusion), visceral metastases (present vs absent) and site. Patients are randomized to 1 of 2 treatment arms.

ELIGIBILITY:
SELECTION OF PATIENTS (MOST IMPORTANT CRITERIA)

Inclusion criteria for first-line therapy

• Histologically confirmed breast cancer with distant metastases

Note:

1. A biopsy from the primary tumor or a metastasis can be used for diagnosis.
2. Patients with non-measurable lesions are eligible.
3. Patients with inoperable, locally advanced breast cancer with lymph node metastases other than ipsilateral locoregional (axillary, infraclavicular, parasternal) or other distant metastases are eligible.
4. Patients with bone metastases with or without bone targeted therapy (bisphosphonates, denosumab) are eligible.
5. Patients with de-novo Stage IV disease are eligible.

   * HER2-positive tumor according to central pathology testing for HER2

Note:

1. A formalin-fixed paraffin-embedded (FFPE) biopsy from the primary tumor or a metastasis has to be used for HER2 status determination. If a biopsy is available from a metastasis, the HER2 testing should be performed using the metastasis.
2. Fine needle aspiration is not acceptable for HER 2 testing. • Women aged ≥18 years

   • WHO performance status 0 to 2
   * Left Ventricular Ejection Fraction (LVEF) ≥50% as determined by either ECHO or MUGA
   * Adequate organ function, evidenced by the following laboratory results:

   Neutrophils >1.5x109/L, platelets >100x109/L, hemoglobin ≥90g/L, total bilirubin ≤1.5xULN (unless the patients has documented Gilbert's disease), AST ≤3xULN, ALT ≤3xULN, AP ≤2.5xULN (except in patients with bone metastases: AP ≤5xULN), creatinine ≤1.5xULN

   Exclusion criteria for first-line therapy

   • Prior chemotherapy for inoperable locally advanced or metastatic breast cancer

   Note:

   Prior neoadjuvant/adjuvant chemotherapy is allowed if doses for anthracyclines have not exceeded 720mg/m2 and 240mg/m2 for epirubicin and doxorubicin, respectively.

   - Re-exposure to paclitaxel is permitted, if the last dose of taxane was given at least 1 year before randomization.

   - Re-exposure to vinorelbine is permitted, if the last dose of vinorelbine was given at least 1 year before randomization.
   * Prior anti-HER2 treatment for metastatic or inoperable breast cancer

   Note:

   Prior neoadjuvant/adjuvant anti-HER2 treatment with trastuzumab and/or lapatinib is allowed.

   • More than one endocrine treatment line for metastatic or inoperable breast cancer exceeding a duration of 1 month

   Note:

<!-- -->

1. Adjuvant endocrine treatment is not counted as one line.
2. Patients progressing on endocrine treatment: this specific endocrine treatment must have been stopped at least 2 weeks prior to randomization.

   • Prior treatment with pertuzumab and/or T-DM1

   • Known leptomeningeal or CNS metastases

   Note:

   A brain MRI or CT scan is mandatory in case of clinical suspicion of CNS metastases.

   • Single bone metastasis treated with radiotherapy (if the bone metastasis is the only tumor lesion)

   Inclusion criteria for second-line therapy • At least one dose of trial therapy in the first-line treatment phase of this trial

   • • Proven disease progression on first-line therapy or radiotherapy of a bone metastasis

   Notes:

   First new parenchymal CNS metastases only do not count as progression requiring the initiation of second line trial treatment. Radiotherapy of a single area only for pain control is allowed and will not count as PD.

   • Adequate organ function, evidenced by the following laboratory results: Neutrophils >1.5x109/L, platelets >100x109/L, hemoglobin ≥90g/L, total bilirubin ≤1.5xULN (unless the patients has documented Gilbert's disease), AST ≤3xULN, AP ≤2.5xULN (except in patients with bone metastases: AP ≤5xULN), creatinine ≤1.5ULN

   • LVEF ≥50% as determined by either ECHO or MUGA

   • QoL questionnaire has been completed.

   Exclusion criteria for second-line therapy

   • Termination of first-line therapy with trastuzumab/pertuzumab due to unacceptable toxicity without objective evidence of disease progression

   • CNS metastases that are untreated, symptomatic, or require therapy to control symptoms, as well as a history of radiation, surgery, or other therapy, including steroids, to control symptoms from CNS metastases within 2 months (60 days) before registration

   • Peripheral neuropathy of CTCAE grade ≥3
   * Interstitial lung disease (ILD) or pneumonitis grade ≥3
   * Any other adverse event which has not recovered to CTCAE grade ≤1 (except alopecia)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2013-03-03 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2020-05-26 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) - Analysis Population: ITT Population 1 | 24 months
  Patients being alive 24 months after randomization. A success is considered if a patient is alive at least 24 months after randomization. Analysis Population: ITT Population 1

SECONDARY OUTCOMES:
OS - Analysis Population: ITT Population 2 | 24 months
  Proportion of patients being alive 24 months after randomization. A success is considered if a patient is alive at least 24 months after randomization. Analysis Population: ITT Population 2
Progression Free Survival (PFS) of first-line treatment ignoring first Central Nervous System (CNS) lesion | 10 / 16 months (PFS will be calculated sustained from randomization until documented PD (ignoring first CNS lesion) or death, whichever occurs first during first-line treatment )
  PFS of first-line treatment ignoring first CNS lesion is the time from randomization to first event progression. A PFS of first-line treatment ignoring first CNS lesion event is defined as (whichever occurs first):
  * Disease progression (PD) after having received first-line treatment and prior to the next treatment
  * Death due to any reason Patients without events will be censored at last tumor assessment date without PFS ignoring first CNS lesion event during the first-line treatment period or prior to starting new treatment.
  Analysis population: ITT Population 1
PFS of second-line treatment | 8 months (PFS will be calculated sustained from registration of second line treatment until documented PD, PD CNS or death, whichever occurs first during second-line treatment)
  PFS of second-line treatment is the time from registration of second-line treatment to progression. A PFS event of second-line treatment is defined as (whichever occurs first):
  * Disease progression after having received second-line treatment and prior to the next treatment
  * PD CNS after having received first-line treatment and prior to the next treatment
  * Death due any reason during the second-line treatment period Patients without events will be censored at last tumor assessment date without PD and PD CNS during the second-line treatment period or prior to starting new treatment.
  Analysis Population: ITT Population 2
PFS of second-line treatment ignoring first CNS lesion | 9 months (PFS will be calculated sustained from registration of second line treatment until documented PD (ignoring first CNS lesion) or death, whichever occurs first during second-line treatment)
  PFS of second-line treatment ignoring first CNS lesion is the time from registration of second-line treatment to the first event occurs. A PFS of second-line treatment ignoring first CNS lesion event is defined as (whichever occurs first):
  * Disease progression after having received second-line treatment and prior to the next treatment
  * Death due any reason during the second-line treatment period Patients without events will be censored at last tumor assessment date without PFS ignoring first CNS lesion event during the second-line treatment period or prior to starting new treatment.
  Analysis Population: ITT Population 2
Time to failure of strategy (TFS) of first- plus second-line treatment | 18 / 24 months (TFS will be calculated sustained from randomization until documented PD, PD CNS or death, whichever occurs first before starting third-line therapy )
  TFS of first plus second-line treatment is the time from randomization to TFS event occurs. A TFS event of first plus second-line treatment is defined as (whichever occurs first):
  * Disease progression after having received the first and second-line treatment and prior to the next treatment
  * PD CNS after having received first- and second-line treatment and prior to the next treatment
  * Death due to tumor prior to the third-line treatment Patients without events will be censored at last tumor assessment without PD and PD CNS during first and second-line treatment period or prior to starting new treatment.
  Analysis Population: ITT Population 1
Overall survival OS | OS will be calculated from randomization until death (estimated median: 32 months)
  OS will be calculated from randomization until death. Patients still alive or lost of follow up are censored at their last date known alive.
  Analysis Population: ITT Population 1
Objective response (OR) of first-line treatment (based on investigator assessment) | 10 / 16 months (OR is defined as the best status of response CR or PR up to first progression or start of a new treatment)
Disease control (DC) of first-line treatment (based on investigator assessment) | 6 months (DC is defined as CR, PR or SD for 6 months after randomization and no PD at 6 month after randomization)
OR of second-line treatment (based on investigator assessment) | 9 months (OR is defined as the best status of response CR or PR after registration for second-line treatment up to second progression or start of a new treatment)
DC of second-line treatment (based on investigator assessment) | 6 months (DC is defined as the response CR, PR or SD for 6 months after registration of second-line treatment)
Adverse events (AEs) according to the NCI CTCAE v4.0 of first-line treatment | Throughout first-line treatment (estimated up to 16 months)
  Adverse events are assessed by the NCI CTCAE v4.0. from registration until registration of second-line treatment or start of follow-up (which occurs first).
AEs according to the NCI CTCAE v4.0 of second-line treatment | Throughout second-line treatment (estimated up to 9 months)
  Adverse events are assessed by the NCI CTCAE v4.0.from second-line registration until PD or start of follow-up (which occurs first) plus 30 days.
AEs grade ≥2 until first progression (ignoring first CNS lesion) | Throughout first-line treatment (estimated up to 16 months)
  Adverse events are assessed by Common terminology criteria for adverse events (CTCAE) v4.0. From randomization until first progression (documented PD, PD CNS or death)
Quality of Life (QoL) | At baseline and every 12 weeks (three-monthly) until progression or up to a maximum of 24 months during 1st line therapy. Within 3 weeks prior to registration, after 12 and 24 weeks during 2nd line therapy.
PFS of third-line treatment | 4 months
  PFS will be calculated sustained from start of third-line treatment to progression (PD, PD CNS or death)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Huober, MD, Study Chair — University of Ulm; Patrik Weder, MD, Study Chair — Cantonal Hospital of St. Gallen; Hervé Bonnefoi, Prof, Study Chair — Institut Bergonié Bordeaux; Epie Boven, MD, Study Chair — Amsterdam UMC, location VUmc
Locations (71):
- France (36):
  - Hopital Sud - Amiens, Amiens
  - ICO - Paul Papin, Angers
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier de Blois, Blois
  - Institut Bergonie, Bordeaux
  - Hôpital Morvan (Brest), Brest
  - Centre Francois Baclesse, Caen
  - Centre Hospitalier Alpes Leman, Contamine-sur-Arve
  - Centre Georges François Leclerc, Dijon
  - Centre Hospitalier de Dracenie, Draguignan
  - Hopital Michallon - Centre Hospitalier Universitaire de Grenoble, Grenoble
  - Clinique Hartmann, Levallois-Perret
  - Centre Oscar Lambret, Lille
  - Chu de Limoges - Hopital Dupuytren, Limoges
  - Centre Hospitalier - Site Hopital du Scorff, Lorient
  - Clinique de la Sauvegarde, Lyon
  - Fondation Hopital Ambroise Pare - Hopital Europeen, Marseille
  - Istitut Paoli Calmettes, Marseille
  - Institut Regional du Cancer Montpellier Val d'Aurelle, Montpellier
  - Centre Azureen de Cancerologie, Mougins
  - Polyclinique de Gentilly, Nancy
  - Centre Catherine de Sienne, Nantes
  - Centre Antoine Lacassagne, Nice
  - Hopital Saint Louis, Paris
  - Centre Hospitalier de Pau, Pau
  - Centre Hospitalier de Perpignan - Hopital Saint Jean, Perpignan
  - Institut Jean Godinot, Reims
  - Clinique Mathilde, Rouen
  - Centre Henri Becquerel, Rouen
  - Curie Site Saint-Cloud, Saint-Cloud
  - ICO - Rene Gauducheau, Saint-Herblain
  - Institut de Cancerologie de la Loire, Saint-Priest-en-Jarez
  - Hopitaux Universitaire de Strasbourg - Hopital Civil, Strasbourg
  - Hopitaux du Leman - Site Georges Pianta, Thonon-les-Bains
  - Institut Claudius Regaud, Toulouse
  - Centre Hospitalier de Valence, Valence
- Universitäts-Frauenklinik Ulm, Ulm, Germany
- Netherlands (13):
  - Almelo_Ziekenhuisgroep Twente, Almelo
  - VUmc University Medical Center, Amsterdam
  - Antoni van Leeuwenhoek / Slotervaart hospital, Amsterdam
  - Reinier de Graaf Gasthuis, Delft
  - Deventer Ziekenhuis, Deventer
  - Catharina Ziekenhuis, Eindhoven
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Leiden_Leids Universitair Medisch Centrum (LUMC), Leiden
  - St. Antonius Ziekenhuis, Ioc Nieuwegein, Nieuwegein
  - St. Franciscus Gasthuis Rotterdam, Rotterdam
  - Vlietland Ziekenhuis, Schiedam
  - Orbis Medisch Centrum, Sittard
  - Haga Ziekenhuis, The Hague
- Switzerland (21):
  - Hirslanden Klinik Aarau, Aarau
  - Kantonspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitaetsspital-Basel, Basel
  - Istituto Oncologico della Svizzera Italiana - Ospedale Regionale Bellinzona e Valli, Bellinzona
  - Inselspital, Bern, Bern
  - RSV-GNW Spitalzentrum Oberwallis, Brig
  - Spitalzentrum Oberwallis, Brig
  - Kantonsspital Graubuenden, Chur
  - Kantonsspital Frauenfeld / Brustzentrum Thurgau, Frauenfeld
  - Hopitaux Universitaires de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois CHUV, Lausanne
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Liestal, Liestal
  - Kantonsspital Luzern, Luzerne
  - Kantonsspital Olten, Olten
  - Kantonsspital St. Gallen, Sankt Gallen
  - Zentrum fuer Tumordiagnostik und Praevention, Sankt Gallen
  - SpitalSTS AG Simmental-Thun-Saanenland, Thun
  - Kantonsspital Winterthur, Winterthur
  - Universitäts Spital Zürich, Zurich

REFERENCES:
- [Derived] Huober J, Weder P, Ribi K, Thurlimann B, Thery JC, Li Q, Vanlemmens L, Guiu S, Brain E, Grenier J, Dalenc F, Levy C, Savoye AM, Muller A, Membrez-Antonioli V, Gerard MA, Lemonnier J, Hawle H, Dietrich D, Boven E, Bonnefoi H; Swiss Group for Clinical Cancer Research, Unicancer Breast Group, and Dutch Breast Cancer Research Group. Pertuzumab Plus Trastuzumab With or Without Chemotherapy Followed by Emtansine in ERBB2-Positive Metastatic Breast Cancer: A Secondary Analysis of a Randomized Clinical Trial. JAMA Oncol. 2023 Oct 1;9(10):1381-1389. doi: 10.1001/jamaoncol.2023.2909. PMID 37561451